CLINICAL TRIAL: NCT00935233
Title: ICICLE- A Study to Investigate the genetiCs of In Situ Carcinoma of the ductaL subtypE
Brief Title: Study of Biomarkers in Blood and/or Tumor Tissue Samples From Patients With Ductal Carcinoma in Situ and From Healthy Volunteers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Queen Mary University of London (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CRUK-ICICLE; CDR0000629681 (Registry Identifier: PDQ (Physician Data Query)); EU-20895
Record Dates: First submitted 2009-07-07; First posted 2009-07-08 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2009-07

CONDITIONS: Breast Cancer
Keywords: ductal breast carcinoma in situ
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating | interventions — Amplified Fragment Length Polymorphism Analysis

INTERVENTIONS:
Genetic: DNA analysis
Genetic: polymorphism analysis
Genetic: protein analysis
Other: laboratory biomarker analysis
Other: questionnaire administration
Other: survey administration

SUMMARY:
RATIONALE: Studying genes in samples of blood and/or tumor tissue from patients with cancer may help doctors identify biomarkers related to cancer.

PURPOSE: This research study is looking at blood and/or tumor tissue samples from patients with ductal carcinoma in situ and blood samples from healthy volunteers.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To collect blood and/or tumor tissue of patients with ductal breast carcinoma in situ (DCIS) and their age- and ethnicity-matched controls to identify the inherited variation that predisposes women to develop DCIS.
* To determine the frequency of these variants.
* To determine the effect of these variants on tumor risk.
* To determine the benefit of testing for these variants in the clinical setting so that those at higher risk could be identified, counseled, and screened.

Secondary

* To analyze the acquired genetic changes within DCIS to identify which cases are more likely to develop invasive disease.

OUTLINE: This is a multicenter study.

All participants complete a questionnaire to collect their family history, a brief medical history, and epidemiological data.

Patients undergo collection of blood and/or tumor tissue samples; DNA is extracted for genotyping, comparison of allele and genotype frequencies (polymorphisms), genetic profiling, DNA analysis, and protein analysis. Histopathology reports are also collected. Healthy volunteers undergo collection of blood samples.

PROJECTED ACCRUAL: A minimum of 3,000 patients and 3,000 controls will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Prior or current diagnosis of pure ductal carcinoma in situ (DCIS)

  * Age ≤ 60 years at the time of diagnosis
  * DCIS with contralateral synchronous or asynchronous invasive breast cancer is permitted
  * DCIS associated with microinvasion (foci < 1 mm) is permitted
* Healthy age- and ethnicity-matched controls

  * No history of DCIS
  * No relative (up to second degree) diagnosed with DCIS

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Collection of blood and/or tumor tissue
Frequency of genetic variants that predispose women to develop ductal carcinoma in situ (DCIS)
Effect of these variants on tumor risk
Benefit of testing for these variants

SECONDARY OUTCOMES:
Analysis of acquired genetic changes within DCIS

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Roylance, MD, Principal Investigator — Barts and the London School of Medicine and Dentistry; Elinor Sawyer, MD — Cancer Research UK
Locations (18):
- United Kingdom (18):
  - North Devon District Hospital, Barnstaple, England
  - Basildon University Hospital, Basildon, England
  - Cumberland Infirmary, Cambridge, England
  - Colchester General Hospital, Colchester, England
  - Dartford & Gravesham NHS Trust, Joyce Green Hospital, Dartford Kent, England
  - Dorset County Hospital, Dorchester, England
  - Northwick Park Hospital, Harrow, England
  - West Middlesex University Hospital, Isleworth, England
  - Barts and the London School of Medicine, London, England
  - Helen Rollason Cancer Care Centre at North Middlesex Hospital, London, England
  - Cancer Research UK Clinical Groups at Guy's King's & St. Thomas' Hospitals, London, England
  - King's College Hospital, London, England
  - Charing Cross Hospital, London, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Princess Royal University Hospital, Orpington, Kent, England
  - Southend University Hospital NHS Foundation Trust, Westcliff-on-Sea, England
  - Dumfries & Galloway Royal Infirmary, Dumfries, Scotland
  - Bronglais District General Hospital, Aberystwyth, Wales